CLINICAL TRIAL: NCT06595069
Title: A Single-Center, Retrospective, Observational Study to Assess the Characteristics and the Real-World Long-Term Effectiveness of Inclisiran in Chinese Adult Patients
Brief Title: A Real-world Study to Assess the Characteristics and Long-term Effectiveness of Inclisiran in Chinese Adult Patients
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: CKJX839A1CN05
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hypercholesterolemia
Keywords: Elevated low-density lipoprotein cholesterol; Inclisiran; Real-world
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Inclisiran Cohort: Chinese adult patients who received at least one treatment with inclisiran.

SUMMARY:
This was a single-center, retrospective, observational study (non-interventional study with secondary use of data) among patients in a real-world setting.

This study used the medical record data from patients in Yiling. Eligible patients who newly initiated inclisiran from 26 January 2022 to 21 August 2023 were included. The retrospective data up to the date of ethics committee approval (April 2024) was collected. The study team collected patient data using an electronic case report form (eCRF) from April 2024 to June 2024.

ELIGIBILITY:
Inclusion criteria:

* Received at least one inclisiran injection during the indexing period.
* Had at least 9 months of follow-up from the index date (had at least one LDL-C assessment during baseline period and at least one LDL-C assessment at 9 months or later).
* Patients signed the informed consent form.

Exclusion criteria:

• Participated in any blinded interventional clinical studies anytime during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Percentage Change From Baseline to Month 9 in Low Density Lipoprotein Cholesterol (LDL-C) Levels | Baseline, Month 9

SECONDARY OUTCOMES:
Absolute Change From Baseline to Month 9 in Low Density Lipoprotein Cholesterol (LDL-C) Levels | Baseline, Month 9
Change From Baseline to Month 9 in Total Cholesterol Levels | Baseline, Month 9
Change From Baseline to Month 9 in Apolipoprotein B Levels | Baseline, Month 9
Change From Baseline to Month 9 in non-High Density Lipoprotein Cholesterol Levels | Baseline, Month 9
Change From Baseline to Month 9 in Serum Apolipoprotein A1 Levels | Baseline, Month 9
Change From Baseline to Month 9 in High Density Lipoprotein Cholesterol Levels | Baseline, Month 9
Change From Baseline to Month 9 in Lipoprotein (a) Levels | Baseline, Month 9
Change From Baseline to Month 9 in Triglyceride Levels | Baseline, Month 9
Number of Patients With at Least two Doses of Inclisiran After the First Injection of Inclisiran | Up to 27 months
Number of Patients who Switched at Least Once From Inclisiran to Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9) Monoclonal Antibody Treatment | Up to 27 months
Number of Patients With Changes in Lipid-lowering Therapies (LLTs) | Up to 27 months
  Changes in LLTs included:
  * LLT dose modification (dose increase, dose decrease).
  * LLT switches.
  * Use of new add-on therapy.
  * LLT interruption.
  * LLT discontinuation.
  * Time between first inclisiran injection and subsequent doses.
Proportion of Days Covered (Adherence) of Inclisiran Over 12 Months | 12 months
  Proportion of Days Covered of inclisiran over 12 months was calculated by the days covered by inclisiran within 12 months divided by 12 months.
Number of Patients per Demographic Category | Baseline
  Demographic categories included:
  * Age
  * Gender
  * Ethnicity
  * Smoking history
  * Alcohol use history
Number of Patients per Clinical Characteristic Category | Baseline
  Clinical characteristics included:
  * Family history of hereditary disease
  * Comorbidities
  * Medication history
  * Concomitant medications and/or therapies
  * Background LLT regimens
Baseline Lipid Levels | Baseline
  Lipids included, but were not limited to, LDL-C, total cholesterol, apolipoprotein B, non-high density lipoprotein cholesterol, serum apolipoprotein A1, high density lipoprotein cholesterol, lipoprotein (a), and triglycerides.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States